CLINICAL TRIAL: NCT06328491
Title: Erdafitinib in Metastatic Steroid-cell Tumor of the Ovary, NOS
Brief Title: Erdafitinib in Metastatic Steroid-cell Ovarian Cancer
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University Health Network, Toronto (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: OZUHN-014; 22-5325 (Other: University Health Network)
Record Dates: First submitted 2022-05-26; First posted 2024-03-25 (Actual); Last update posted 2024-03-25 (Actual); Status verified 2024-03

CONDITIONS: Ovarian Cancer; Steroid Cell Tumor, Malignant
MeSH Terms: conditions — Ovarian Neoplasms | interventions — erdafitinib

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Erdafitinib in metastatic steroid-cell tumor of the ovary (Experimental): Erdafitinib, 8 mg, orally, once daily. Dose increase to 9 mg once daily may be considered based on serum phosphate levels and tolerability.
  Interventions: Drug: Erdafitinib

INTERVENTIONS:
Drug: Erdafitinib — Protein Kinase Inhibitor
  Other Names: Balversa

SUMMARY:
This is a single participant study of erdafitinib for the treatment of a patient with metastatic steroid-cell tumor of the ovary.

DETAILED DESCRIPTION:
Erdafitinib was approved by FDA in 2019 for patients with locally advanced or metastatic urothelial carcinoma with susceptible FGFR alterations. Blocking the FGF/FGFR signaling axis by tyrosine kinase inhibitors was proved to be a successful therapeutic strategy in numerous tumor types. Erdafitinib was the first approved FGFR-TKI for treating metastatic urothelial carcinoma based on remarkable results of the phase II trial (BLC2001), that enrolled 212 patients of whom 101 patients was treated with uptitration dose of 9mg daily. The median follow-up for efficacy was 24 months (IQR 22.7*26.6). The objective response rate was 40% (95% CI) of 101 patients of uptitration group. The common grade 3-4 adverse events were stomatitis and hyponatremia4. A phase III trial (NCT03390504) is being performed to compare the efficacy of Erdafitinib versus Vinflunine or Docetaxel or Pembrolizumab in advanced urothelial cancer. Multiple clinical trials are being conducted on the effectiveness of Erdafitinib in a variety of cancers that harbors FGFR alterations. These indicate the potential to improve control in this rare disease which otherwise is devastating and associated with a very high likelihood of recurrence and poor survival.

ELIGIBILITY:
Inclusion Criteria & Exclusion Criteria:

This is a single patient study and the protocol was specifically designed for this single patient. This patient case was discussed in the hospital expert molecular tumor board rounds consisting of representatives from specialist genomic profiling and gynecologic medical oncology departments. The discussion surrounded the best next therapeutic option in this extremely rare cancer subtype without clear standard of care guidelines. The recommendation from this discussion was to perform radiation therapy to her bone lesion and access target treatment against FGFR4 amplification, such as Erdafitinib that is a pan FGFR kinase inhibitor and binds to and inhibits FGFR1, FGFR2, FGFR3, and FGFR4 enzyme activity.

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 1 (Actual)
Dates: Start 2022-05-30 (Actual); Primary Completion 2022-08-22 (Actual); Study Completion 2022-08-22 (Actual)

PRIMARY OUTCOMES:
Tumor response | Until disease progression or until the investigator deems that it is in the patient's best interest to stop study treatment whichever came first, assessed up to 3 months.
  Response will be measured radiographically with restaging CT thorax, abdomen and pelvis every 9-12 weeks while on treatment.
Overall health status | Until disease progression or until the investigator deems that it is in the patient's best interest to stop study treatment whichever came first, assessed up to 3 months.
  Clinical endpoints will include overall performance status including Eastern Cooperative Oncology Group (ECOG) score and patient-reported symptoms. There will be no formal data analysis.

CONTACTS AND LOCATIONS:
Overall Officials: Amit Oza, M.D., Principal Investigator — Princess Margaret Cancer Centre
Locations (1):
- Princess Margaret Cancer Centre, Toronto, Ontario, Canada